CLINICAL TRIAL: NCT03604614
Title: A Randomized Controlled Clinical Trial of Hyperthermic Intraperitoneal Chemotherapy for Advanced Gastric Cancer With Peritoneal Metastatis
Brief Title: Hyperthermic Intraperitoneal Chemotherapy for Advanced Gastric Cancer With Peritoneal Metastatis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangdong Provincial Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Wei Wang, Wei Wang M.D., PhD.，Head of Gastroenterology, Principal Investigator, Clinical Professor, Guangdong Provincial Hospital of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GDPHCM-GI-03
Record Dates: First submitted 2018-06-14; First posted 2018-07-27 (Actual); Last update posted 2018-07-27 (Actual); Status verified 2018-07

CONDITIONS: Stage IV Gastric Cancer With Metastasis; Hyperthermic Intraperitoneal Chemotherapy; Exploratory Behavior
Keywords: peritoneal metastatis; Hyperthermic Intraperitoneal Chemotherapy; Advanced gastric adenocarcinoma
MeSH Terms: conditions — Exploratory Behavior | interventions — Hyperthermic Intraperitoneal Chemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIPEC and chemotherapy (Experimental): Hyperthermic Intraperitoneal Chemotherapy and SOX（Tiggio+Oxaliplatin ）
  Interventions: Drug: Hyperthermic Intraperitoneal Chemotherapy
- Without HIPEC (Sham Comparator): Without Hyperthermic Intraperitoneal Chemotherapy，Only SOX（Tiggio+Oxaliplatin ）
  Interventions: Drug: Without Hyperthermic Intraperitoneal Chemotherapy

INTERVENTIONS:
Drug: Hyperthermic Intraperitoneal Chemotherapy — The investigators use Paclitaxel as peritoneal hyperthermic perfusion chemotherapy drugs，75mg/m2 for the first time，50mg/m2 for the second time and third time.The chemotherapy is SOX(Tiggio d1-d14 bid po and Oxaliplatin 130mg/m2 ivd d1 qd).The Tiggio dosage depends on the patient's body surface area, body surface area <1.25m2 40mg/time, 1.25-1.50m2 50mg/time, >1.50m2 60mg/time.
  Arms: HIPEC and chemotherapy
Drug: Without Hyperthermic Intraperitoneal Chemotherapy — The chemotherapy is SOX(Tiggio d1-d14 bid po and Oxaliplatin 130mg/m2 ivd d1 qd).The Tiggio dosage depends on the patient's body surface area, body surface area <1.25m2 40mg/time, 1.25-1.50m2 50mg/time, >1.50m2 60mg/time.
  Arms: Without HIPEC

SUMMARY:
The incidence rate of gastric cancer is high in Southeast Asia, so is the mortality rate.Due to the lack of specific performance, about 5%-20% of patients have found peritoneal metastases at the time of first diagnosis.At present, clinical studies on HIPEC in the treatment of patients with advanced gastric cancer peritoneal metastasis are almost related to abdominal perfusion after laparoscopic gastrectomy.Herein, we conduct a single-centre randomized controlled trial to explore the safety and feasibility of laparoscopic exploration combined with HIPEC in the treatment of advanced gastric cancer with peritoneal metastasis.

DETAILED DESCRIPTION:
Gastric cancer is one of the most common digestive tumors in the world.In China, advanced gastric cancer with severe local progression or distant metastasis is more common.Gastric cancer with peritoneal carcinomatosis has an extremely poor prognosis,with a median survival of less than 6 months.Hyperthermic Intraperitoneal Chemotherapy (HIPEC) is currently a treatment for malignant tumors in the abdominal cavity and prevents tumor recurrence and metastasis.Studies have shown that hyperthermic intraperitoneal perfusion chemotherapy (HIPEC) has good clinical efficacy in the prevention and treatment of peritoneal metastasis of gastric cancer and its associated malignant ascites.Therefore,we conduct a single-centre randomized controlled trial to explore the safety and feasibility of HIPEC in the treatment of advanced gastric cancer with peritoneal metastasis. The metahnism of HIPEC is taking advantage of the difference in temperature sensitivity between cancer cells and normal cells. Perfusion of the abdominal cavity with a chemical fluid of the appropriate temperature can be performed. Suitable high temperatures can directly kill tumor cells.It is generally believed that the optimal temperature for the treatment of tumors is 42.5°C to 44°C.In this study,we set the temperature 43°C. Paclitaxel is a novel broad-spectrum antitumor drug,which has a unique anti-cancer mechanism.We use Paclitaxel as peritoneal hyperthermic perfusion chemotherapy drugs.The chemotherapy is SOX(Teggio and Oxaliplatin),.The primary endpoint is PFS. Secondary endpoints are one-year OS、canversion rate and ascites assessment. A phase III study PHOENIX-GC trial had finished enrollment,and the conclusion was the median OS 17.7 and 15.2 months respectively for IP and SP.The primary analysis did not show the statistical superiority of the IP regimen.The sensitivity analysis IP considering the imbalance of ascites, suggested clinical efficacy of IP PTX in gastric cancer with peritoneal metastasis. For this reason,we conduct a trial to explore the safety and feasibility of HIPEC in the treatment of advanced gastric cancer with peritoneal metastasis.

ELIGIBILITY:
Inclusion Criteria:

* Primary gastric adenocarcinoma diagnosed pathologically by endoscopic biopsy；
* Laparoscopic exploration of patients with advanced gastric adenocarcinoma of peritoneal metastasis；
* Eastern Cooperative Oncology Group (ECOG): 0 ot 1；
* American Society of Anesthesiologists （ASA） score: I to Ⅲ；
* Patient informed consent。

Exclusion Criteria:

* Pregnancy or female in suckling period；
* Severe mental illness；
* Preoperative imaging or intraoperative exploration reveals distant blood, liver, lung, and brain metastases；
* 5 years of history of other malignant diseases；
* A history of unstable angina or myocardial infarction within 6 months；
* History of cerebral infarction or cerebral hemorrhage within 6 months；
* A history of sustained systemic corticosteroid treatment within 1 month；
* Emergency operation due to complication (bleeding, perforation or obstruction) caused by primary tumor；
* Pulmonary function test FEV1 <predicted value 50%。

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2017-08-24 (Actual); Study Completion 2020-08-24 (Estimated)

PRIMARY OUTCOMES:
PFS | From date of randomization until the date of first documented progression or date of death for tumor cause, whichever came first, assessed 7 months
  Progression-free survival

SECONDARY OUTCOMES:
1-year survival | one year
  1-year overall survival rate
Ascites assessment | Intraoperative
  Ascites assessment during surgery
Median survival | From date of randomization until only 50% of individuals living for tumor cause, assessed 2 years
  Median Survival Time

CONTACTS AND LOCATIONS:
Overall Officials: Wei Wang, Principal Investigator — Guangdong Provincial Hospital of Traditional Chinese Medicine; Wenjun Xiong, Principal Investigator — Guangdong Provincial Hospital of Traditional Chinese Medicine
Locations (1):
- Guangdong Province Hospital of Chinese Medicine, the Second Affiliated Hospital of Guangzhou University of Chinese Medicine, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
The data has not been published.

REFERENCES:
- [Derived] Luo L, Zhang Z, Zeng H, Xu Y, Peng Y, Huang H, Lin Z, Xiong W, Wang W. Hyperthermic intraperitoneal chemotherapy plus SOX chemotherapy versus SOX chemotherapy alone in patients with gastric cancer and peritoneal metastasis: a phase II randomized clinical trial. J Gastrointest Oncol. 2025 Feb 28;16(1):17-26. doi: 10.21037/jgo-24-807. Epub 2025 Jan 9. PMID 40115934